CLINICAL TRIAL: NCT00312455
Title: Cholesterol and Fatty Acids in Cocaine Addiction Relapse
Brief Title: Effects of Fatty Acid Supplementation on Substance Dependent Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Laure Buydens-Branchey, MD, VA New York Harbor Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA015360-03 (NIH); DPMC
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Substance-related Disorders
Keywords: Substance abuse; Depression; Aggression
MeSH Terms: conditions — Substance-Related Disorders; Depression; Aggression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug Treatment
  Interventions: Drug: Pro-eicosapentaenoic acid (EPA); Drug: Pro-docosapentaenoic acid (DPA)
- 2 (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pro-eicosapentaenoic acid (EPA) — 450 mg 5x/day
  Arms: 1
Drug: Pro-docosapentaenoic acid (DPA) — 100mg 5x/day
  Arms: 1
Drug: Placebo — 5 capsules/day
  Arms: 2

SUMMARY:
Many substance dependent individuals continue to abuse a variety of substances during treatment for their disorder. Often, substance dependent individuals are co-diagnosed with depression and violence problems. Supplements of n-3 polyunsaturated fatty acids (PUFAs) may play a role in treating individuals with such substance abuse problems. The purpose of this study is to evaluate the effectiveness of the n-3 PUFAs eicosapentaenoic acid (EPA) and docosapentaenoic acid (DPA) in treating relapse, aggression, and depression in substance dependent individuals.

DETAILED DESCRIPTION:
Past research suggests that low levels of some PUFAs play a role in the pathophysiology of depressive and aggressive disorders. In addition, there is also evidence that PUFAs play a role in treating substance dependent individuals. The purpose of this study is to determine the efficacy of EFA and DPA in treating substance dependent individuals.

Participants will be randomly assigned to receive either 3 grams of n-3 PUFAs or placebo. Treatment will last 3 months, followed by an observation period of 3 months. Study visits will occur monthly and will last approximately one hour. Study visits will include blood tests and a physical exam. Throughout the study, participants will continue to receive standard substance abuse treatment and will complete urine tests at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Current or history of drug or alcohol dependence
* Used substances of abuse during the 3 months prior to study entry
* Enrolled in one of the VA New York Harbor Healthcare System Brooklyn campus substance abuse clinics

Exclusion Criteria:

* Current or history of hallucinations, delusions, or memory problems
* Major physical illness (e.g., cardiovascular, pulmonary, gastrointestinal, renal, neuromuscular, or endocrine disorder)
* Liver function test greater than one standard deviation above upper normal limit
* Allergic to fish

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laure Buydens-Branchey, MD, Principal Investigator — VA New York Harbor Healthcare System